CLINICAL TRIAL: NCT04835324
Title: Regorafenib Treatment Patterns and Survival Outcomes in Advanced Colorectal Cancer: A Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Beijing Hospital (Other Government); Jiangsu Cancer Institute & Hospital (Other); The Affiliated Hospital of Qingdao University (Other); Shanxi Province Cancer Hospital (Other); Affiliated Hospital of Hebei University (Other); Shandong Cancer Hospital and Institute (Other); The First Affiliated Hospital of Zhengzhou University (Other); Hebei Medical University Fourth Hospital (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Chief Physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: ChineseAcademyMedicalSciences
Record Dates: First submitted 2021-03-28; First posted 2021-04-08 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

SUMMARY:
This is a multi-center, retrospective, real-world study. The purpose of this study is to observe the effectiveness and safety of regorafenib in Chinese advanced colorectal cancer patients.

The main observational goals include overall survival(OS), 6 month OS rate, 1 year OS rate, and treatment time failure (TTF), other study goals include objective response rate( ORR)、Disease control rate（DCR）and adverse event(AE) of regorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer confirmed by pathological tissue or cytology；
2. The pathological type of colorectal tumor was adenocarcinoma；
3. Patients with recurrent or metastatic, unresectable advanced colorectal cancer；
4. Patients who received regorafenib at least one period treatment.

Exclusion Criteria:

1. Patients participating in other interventional clinical studies while taking regorafenib;
2. Patients with other malignant tumors within 5 years before regorafenib treatment, except for cured cervical carcinoma in situ, skin squamous cell carcinoma or basal cell carcinoma, early papillary thyroid carcinoma, etc.;
3. The investigator deems that there are other factors that are not suitable for patients who participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About 1000 patients in this observational study were recruited in 10 Chinese medical centers since July 2017 to October 2020.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
6-month Overall Survival rate | 6 month
  6 months OS rate of patients who received regorafenib treatment.
1 year Overall Survival rate | 1 year
  1 year OS rate of patients who received regorafenib treatment.
overall survival | 1 year
  overall survival of patients who received regorafenib treatment.

SECONDARY OUTCOMES:
objective response rate | 1 year
  Investigator assessed according to RECIST v1.1
Disease control rate | 1 year
  Investigator assessed according to RECIST v1.1
Incidence of Adverse Events (AEs) | 1 year
  Number of patients with AE, treatment-related AE (TRAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Yunbo Zhao, Study Chair — Beijing Hospital; Liangjun Zhu, Study Chair — Jiangsu Cancer Institute & Hospital; Zimin Liu, Study Chair — The Affiliated Hospital of Qingdao University; Wei Bai, Study Chair — Shanxi Provincial Cancer Hospital; Aimin Zang, Study Chair — Affiliated Hospital of Hebei University; Bo Liu, Study Chair — Shandong Cancer Hospital and Institute; Hong Zong, Study Chair — The First Affiliated Hospital of Zhengzhou University; Shengmian Li, Study Chair — The fourth hospital of Hebei medical university and hebei cancer hospital; Xiujuan Qu, Study Chair — First Hospital of China Medical University; Aiping Zhou, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (2):
- China (2):
  - Cancer Hospital,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing

REFERENCES:
- [Derived] Qu W, Liu Z, Chen X, Liu B, Zhao Y, Yan H, Qu X, Li S, Zang A, Sun Y, Zhu L, Zhou A. Regorafenib monotherapy or combined with an immune-checkpoint inhibitor as later-line treatment for metastatic colorectal cancer: a multicenter, real-world retrospective study in China. BMC Cancer. 2024 Jan 2;24(1):22. doi: 10.1186/s12885-023-11700-w. PMID 38166647